CLINICAL TRIAL: NCT00477178
Title: The Effect of Codeine on Driving Abilities
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Borchgrevink, Petter C, Norwegian University of Science and Technology
Other Study IDs: 133-04REK
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2007-05

CONDITIONS: Healthy
Keywords: possible problems using codeine when driving

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- chronic non-malignant pain codeine: patients having chronic non-malignant pain, living in Trondheim or the four adjacent counties and treated at the Center for Pain and Complex Disorders at St. Olav University Hospital - on long-term codeine therapy
- chronic non-malignant pain: patients having chronic non-malignant pain, living in Trondheim or the four adjacent counties and treated at the Center for Pain and Complex Disorders at St. Olav University Hospital - NOT on long-term codeine therapy
- healthy: healthy controls

SUMMARY:
20 chronic pain patients using codeine are compared with 20 chronic patients not using opioids and 20 healthy volunteers with respect to driving ability measured by neurophysiological tests and driving in a car simulator.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic pain
* driving more than 50 000 km

Exclusion Criteria:

* addiction
* eyesight disorders

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: chronic pain patients driving more than 50,000 km/yr
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2004-08; Primary Completion 2005-05 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petter C Borchgrevink, Professor, Study Chair — Norwegian University of Science and Technology

REFERENCES:
- [Result] Nilsen HK, Landro NI, Kaasa S, Jenssen GD, Fayers P, Borchgrevink PC. Driving functions in a video simulator in chronic non-malignant pain patients using and not using codeine. Eur J Pain. 2011 Apr;15(4):409-15. doi: 10.1016/j.ejpain.2010.09.008. Epub 2010 Oct 13. PMID 20947399